CLINICAL TRIAL: NCT06190639
Title: A Clinical Study of Sintilimab as Adjuvant Therapy in Node-positive Esophageal Squamous Cell Carcinoma After Radical Surgery Without Neoadjuvant Therapy
Brief Title: A Clinical Study of Sintilimab as Adjuvant Therapy in Node-positive ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Changchun Wang, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-768
Record Dates: First submitted 2023-12-09; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: sintilimab

INTERVENTIONS:
Drug: sintilimab — 200 mg once on day 1, every 21 days

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of sintilimab as adjuvant therapy in node-positive esophageal squamous cell carcinoma after radical surgery without neoadjuvant therapy. The main question it aims to answer is:

• Efficacy of sintilimab as adjuvant therapy Participants will receive sintilimab 200 mg once on day 1, every 21 days(Q3W).

ELIGIBILITY:
Inclusion Criteria:

1. Signed an Informed Consent Form
2. Participant type and target disease characteristics:

   * ECOG PS 0-1
   * Histologically confirmed T1-3N+M0 thoracic esophageal squamous cell cancer (AJCC 8th)
   * can tolerate radical resection of esophageal cancer
   * Resection must be performed within 4-12 weeks prior to enrollment
   * All participants must be confirmed disease-free by physical and imaging examinations within 4 weeks prior to enrollment. Imaging examinations must include CT/MRI scans of the neck, chest and abdomen.
   * All baseline laboratory tests will be evaluated as required and results should be available within 28 days prior to enrollment. Laboratory test values must be selected according to the following criteria (CTCAE V5.0):

     1. WBC ≥2000/μL;
     2. Neutrophils ≥1500/μL;
     3. Platelets ≥100 x 103/μL;
     4. Hemoglobin ≥9.0 g/dL;
     5. Creatinine: Serum creatinine ≤1.5 x above normal (ULN) or creatinine removal rate > 50mL/ min (Cockcroft/Gault formula);
     6. AST ≤3 x ULN;
     7. ALT ≤3 x ULN;
     8. Total bilirubin ≤1.5 x ULN (except for subjects with Gilbert syndrome, where total bilirubin must be < 3 x ULN);
3. Age and fertility status:

   * Age ≥18 years old
   * Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity of HCG is 25 IU/L or equivalent) within 24 hours before starting study treatment.
   * Women must be non-breastfeeding

Exclusion Criteria:

1. Target disease

   * The presence of locally advanced unresectable (regardless of stage) or metastatic disease.
   * Cervical and abdominal esophageal tumors.
2. Medical history and concurrent diseases

   * Complete resection followed by treatment for the removed esophageal cancer (e.g., chemotherapy, targeted drugs, radiation, or biotherapy).
   * Participants with ≥ grade 2 peripheral neuropathy
   * Participants with active, known, or suspected autoimmune diseases. Participants with type I diabetes, hypothyroidism requiring only hormone replacement therapy, skin conditions that do not require systemic treatment (such as vitiligo, psoriasis, or hair loss), or conditions that are not expected to recur without external irritants, may be enrolled.
   * Glucocorticoids are required for 14 days prior to treatment (daily>10 mg equivalent dose of prednisone) or other immunosuppressive drugs for systemic treatment.

   If there is no active autoimmune disease, inhaled or topical steroid hormones are permitted, and daily>10 mg prednisone equivalent dose of adrenal hormone replacement therapy.
   * A known history of testing positive for human immunodeficiency virus (HIV) or a known history of acquired immunodeficiency syndrome (AIDS)
   * Participants with a serious or uncontrolled medical condition.
   * Radiotherapy, chemotherapy, immunotherapy, esophagectomy, esophagus-gastric junction, and gastric surgery were performed before the trial.
   * Participants with severe cardiovascular or pulmonary disease, interstitial pneumonia, or a history of prior interstitial pneumonia.
   * Active malignancy within the last 3 years, other than locally curable cancers that have apparently been cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
   * Participants with a serious or uncontrolled medical condition
3. Physical and laboratory examination

   * Participants were found to have active hepatitis B (Hepatitis B surface antigen [HBsAg] positive or hepatitis C virus (HCV) positive (HCV RNA positive) Sex). Participants with prior HBV infection or recovered HBV infection (defined as having hepatitis B core antibodies [HBcAb] and no HBsAg) were eligible. HBV DNA must be obtained from these patients before treatment. Participants who are HBV carriers or require antiviral therapy are not eligible to participate. Participants who were positive for HCV antibodies were eligible only if the PCR for HCV RNA was negative.
4. Allergies and adverse drug reactions

   * History of allergy or hypersensitivity to study drug ingredients.
   * A history of severe hypersensitivity to any monoclonal antibody.
5. Other exclusion criteria

   * Participants who do not understand or may not comply with the requirements of the trial
   * Participants had an active infection requiring systemic treatment in the 28 days prior to first dosing
   * Some obvious diseases that the researchers believe should be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | assessed up to 36months
  From date of randomization until the date of first documented progression

SECONDARY OUTCOMES:
Overall survival (OS) | assessed up to 60 months
  From date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China